CLINICAL TRIAL: NCT05949593
Title: PHase 3, Multicenter, RandOmized, Double-masked, PlacEbo-CoNtrolled Study of TInlarebant to EXplore Safety and Efficacy in the Treatment of Geographic Atrophy (the PHOENIX Study)
Brief Title: Phase 3, Randomized, Placebo-Controlled Study of Tinlarebant to Explore Safety and Efficacy in Geographic Atrophy
Acronym: PHOENIX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Belite Bio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LBS-008-CT05
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Geographic Atrophy
Keywords: LBS-008; Tinlarebant; GA
MeSH Terms: conditions — Geographic Atrophy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Eligible subjects will be randomly assigned to begin treatment in 2:1 ratio to receive the study drug (either Tinlarebant 5 mg or matching placebo)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LBS-008, Tinlarebant (Experimental)
  Interventions: Drug: Tinlarebant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tinlarebant — 5 mg tablet taken orally once a day
  Arms: LBS-008, Tinlarebant
Drug: Placebo — Placebo tablets for tinlarebant 5 mg prepared similarly.
  Arms: Placebo

SUMMARY:
This Phase 3, multicenter, double-masked, parallel-group, placebo-controlled, randomized, fixed-dose clinical study is designed to evaluate the efficacy and safety of tinlarebant (LBS-008) in subjects diagnosed with GA.

DETAILED DESCRIPTION:
Subjects will be randomized in a 2:1 ratio to receive either tinlarebant or placebo. The study treatment will be administered orally once daily from baseline (Day 1) through the final day of Month 24.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a confirmed diagnosis of GA with atrophic lesions in 1 or both eyes.
* Minimum BCVA is required in the study eye

Exclusion Criteria:

* The presence of diabetic macular edema or macular disease in either eye.
* Diabetic retinopathy more advanced than mild nonproliferative diabetic retinopathy, or any other retinal vascular disease in either eye.
* Uncontrolled diagnosed glaucoma in the study eye

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 429 (Estimated)
Dates: Start 2023-07-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
To measure the rate of change (growth rate slope) in geographic atrophy (GA) lesion size | From baseline to Month 24]

SECONDARY OUTCOMES:
To measure the change in best-corrected visual acuity (BCVA) as assessed using the Early Treatment Diabetic Retinopathy Study (ETDRS) scale | From baseline to Month 24
To measure changes in the area and size of the inner/outer segment junction of photoreceptors by spectral domain optical coherence tomography (SD-OCT) | From baseline to Month 24

CONTACTS AND LOCATIONS:
Locations (47):
- United States (22):
  - Belite Study Site, Phoenix, Arizona
  - Belite Study Site, Arcadia, California
  - Belite Study Site, Beverly Hills, California
  - Belite Study Site, Huntington Beach, California
  - Belite Study Site, Los Angeles, California
  - Belite Study Site, Palo Alto, California
  - Belite Study Site, San Diego, California
  - Belite Study Site, Lakeland, Florida
  - Belite Study Site, Hagerstown, Maryland
  - Belite Study Site, Saint Louis Park, Minnesota
  - Belite Study Site, Westbury, New York
  - Belite Study Site, Cary, North Carolina
  - Belite Study Site, Durham, North Carolina
  - Belite Study Site, Wake Forest, North Carolina
  - Belite Study Site, Portland, Oregon
  - Belite Study Site, Philadelphia, Pennsylvania
  - Belite Study Site, Sewickley, Pennsylvania
  - Belite Study Site, Germantown, Tennessee
  - Belite Study Site, Abilene, Texas
  - Belite Study Site, Dallas, Texas
  - Belite Study Site, San Antonio, Texas
  - Belite Study Site, Warrenton, Virginia
- Australia (6):
  - Belite Study Site, Chatswood, New South Wales
  - Belite Study Site, Strathfield, New South Wales
  - Belite Study Site, Brisbane, Queensland
  - Belite Study Site, Adelaide, South Australia
  - Belite Study Site, East Melbourne, Victoria
  - Belite Study Site, Crawley, Western Australia
- China (5):
  - Belite Study Site, Beijing, Beijing Municipality
  - Belite Study Site, Chengdu, Sichuan
  - Belite Study Site, Beijing
  - Belite Study Site, Guandong
  - Belite Study Site, Zhejiang
- Czechia (2):
  - Belite Study Site, Ostrava
  - Belite Study Site, Prague
- France (4):
  - Belite Study Site, Dijon
  - Belite Study Site, Écully
  - Belite Study Site, Lyon
  - Belite Study Site, Marseille
- Switzerland (2):
  - Belite Study Site, Basel
  - Belite Study Site, Lausanne
- Taiwan (3):
  - Belite Study Site, Taichung
  - Belite Study Site, Taipei
  - Belite Study Site, Taoyuan District
- United Kingdom (3):
  - Belite Study Site, Great Yarmouth
  - Belite Study Site, Harrow
  - Belite Study Site, London

IPD SHARING:
Plan to Share IPD: No